CLINICAL TRIAL: NCT01708447
Title: Feasibility Study: Evaluation of the Efficacy of a Liposome-encapsulated Lidocaine Topical Anesthetic for Reducing Discomfort Associated With Ultherapy™ Treatment
Brief Title: Feasibility Study: Evaluate the Effectiveness of Using a Topical Anesthetic Prior to Ultherapy™ Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ULT-117
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2013-06

CONDITIONS: Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical anesthetic - L.M.X.4.® cream (Active Comparator): Topical anesthetic cream, L.M.X.4.® cream, applied to one side of the face and neck prior to Ulthera System treatment.
  Interventions: Drug: L.M.X.4.® cream; Device: Ulthera System Treatment
- Placebo cream (Placebo Comparator): A placebo cream with similar consistency and color will be applied to the other side of the face and neck prior to Ulthera System treatment.
  Interventions: Other: A placebo cream; Device: Ulthera System Treatment

INTERVENTIONS:
Drug: L.M.X.4.® cream — A lidocaine topical anesthetic cream
  Other Names: A lidocaine topical anesthetic cream
  Arms: Topical anesthetic - L.M.X.4.® cream
Other: A placebo cream — Placebo cream containing no anesthetic properties.
  Arms: Placebo cream
Device: Ulthera System Treatment — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.; Ultrasound treatment for skin tightening

SUMMARY:
This study will evaluate the efficacy of a lidocaine topical anesthetic (numbing cream) for reducing discomfort associated with Ultherapy™ treatment.

DETAILED DESCRIPTION:
All subjects will receive a full face and neck Ultherapy™ treatment. Thirty (30) minutes prior to treatment, a topical anesthetic (numbing cream) will be applied to one side of the face and neck and a placebo cream with similar consistency and color will be applied to the other side of the face and neck, in a randomized fashion. The subject and investigator or sub-investigator performing Ultherapy™ treatment will be blinded to the side to which the topical anesthetic is applied. Pain scores will be collected following treatment of each section of the face and neck on both sides. Subjects will return for a 90-day post-treatment visit to assess improvement in skin laxity, and overall lifting and tightening of skin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 30 to 65 years.
* Chosen an Ultherapy™ treatment as part of their treatment regimen.
* Subject in good health.
* Skin laxity on the face and neck.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the followup period.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study

Exclusion Criteria:

* Known sensitivity to lidocaine or any other anesthetic of the amide type.
* History of anaphylactic shock.
* Presence of an active systemic or local skin disease that may affect wound healing.
* Current therapy with class I antiarrhythmic drugs (e.g., tocainide, mexiletine).
* Known or suspected hypersensitivity to LMX-4 active substance, or any of the amide-type local anaesthetics, or any of the excipients (protocol section 10.3).
* Severe solar elastosis.
* Excessive subcutaneous fat in the face and neck.
* Body mass index of 30 or greater.
* Excessive skin laxity on the face and neck.
* Significant scarring in areas to be treated.
* Significant open facial wounds or lesions.
* Severe or cystic acne on the face.
* Presence of a metal stent or implant in the facial area to be treated.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Treatment-related pain | During treatment
  The validated 10-point pain NRS scale will be used to measure average pain scores reported by subject immediately after each facial region is treated.

SECONDARY OUTCOMES:
Improvement in skin laxity. | 90 days post-treatment
  Improvement in overall lifting and tightening of skin as determined by a masked, qualitative assessment of photographs.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Gitt, MD, Principal Investigator — North Valley Plastic Surgery
Locations (1):
- North Valley Plastic Surgery, Phoenix, Arizona, United States